CLINICAL TRIAL: NCT00785057
Title: A Retrospective, Multi Centre, Non-interventional, Observational Study to Compare Treatment Pattern and Factors That Affect BP Control in Patients With and Without Stroke
Brief Title: Retrospective Treatment Pattern Survey for the Patient With and Without History of Stroke
Acronym: SAPIENCE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-CKR-DUM-2008/4
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension
Keywords: Hypertension; Stroke; Neurology; JNC7; 2007 ESH-ESC guidelines; survey
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Hypertension patients with history of stroke
- 2: Hypertension patients without history of stroke

SUMMARY:
This study will compare hypertension treatment pattern of stroke patients with non-stroke patients receiving medical care from outpatient clinics at neurology specialty centers in Korea. It will evaluate target BP achievement rate in patients with stroke compared to patients without stroke and investigate factors affecting BP target goal efficacy in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients attending neurology specialty centers, either with or without history of stroke, receiving hypertension medication

Exclusion Criteria:

* Secondary hypertension patients
* Patients not receiving hypertension medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension outpatients coming to the Neurology Department
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure, History of stroke, Antihypertensive medication | After collecting all Patient Record Form.

SECONDARY OUTCOMES:
Blood pressure, History of stroke, antihypertensive medication, Classification of stroke, Risk factors, Concomitant medication, etc. | After collecting all Patient Record Form.

CONTACTS AND LOCATIONS:
Overall Officials: Joonwoo Bahn, Study Director — Astrazenca Korea medical dept.
Locations (8):
- South Korea (8):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Sungnam, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Deagu
  - Research Site, Deajeon
  - Research Site, Kwangju
  - Research Site, Seoul